CLINICAL TRIAL: NCT03832361
Title: A Phase II Evaluation of the Safety and Efficacy of Mirvetuximab Soravtansine (IMGN853) in Women With Folate Receptor-α Positive Persistent or Recurrent Endometrial Cancer
Brief Title: Evaluation of Mirvetuximab Soravtansine (IMGN853) in Women With Folate Receptor-α Positive Endometrial Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alessandro Santin (Other)
Collaborators: ImmunoGen, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Alessandro Santin, Professor of Obstetrics, Gynecology, and Reproductive Sciences, Yale University
Organization: Yale University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000023841
Record Dates: First submitted 2019-02-04; First posted 2019-02-06 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — mirvetuximab soravtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IMGN853 (Experimental): IMGN853 administered 6 mg/kg adjusted ideal body weight (AIBW) once every three weeks (Q3W)
  Interventions: Drug: IMGN853

INTERVENTIONS:
Drug: IMGN853 — IMGN853 6 mg/kg intravenously every 3 weeks until disease progression
  Other Names: mirvetuximab soravtansine

SUMMARY:
The purpose of this study is to evaluate the activity and safety profile of mirvetuximab soravtansine (IMGN853) in patients with type II endometrial cancers that overexpress folate receptor alpha (FRα).

DETAILED DESCRIPTION:
This study will enroll patients with persistent or recurrent FRα-positive uterine serous carcinoma (pure or mixed), Grade 3 endometrial adenocarcinoma, or carcinosarcoma with high grade serous or Grade 3 endometrioid components. All patients must have measurable disease. The primary objective of the study is to assess the activity of IMGN853 as measured by objective response rate (ORR). The secondary objectives are to assess the duration of overall survival (OS), progression-free survival (PFS) and durable disease control rate (DDCR), as well as the safety profile of IMGN853 in endometrial carcinoma patients. Exploratory/correlative objectives are to correlate ORR, PFS, and OS with the level of folate receptor α expression and explore use of circulating tumor (ct) DNA as a biomarker for disease response and compare its performance to cancer antigen 125 (CA-125). All enrolled patients will receive IMGN853 at a dose of 6 mg/kg administered intravenously once every 3 weeks until unacceptable toxicity or progression of disease requiring discontinuation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Radiologically confirmed (ie, CT scan and/or MRI) persistent or recurrent endometrial cancer
* Patients must have one of the following pathologically documented, definitively diagnosed tumor types: Uterine serous carcinoma (Pure or Mixed), Grade 2 or Grade 3 endometrial adenocarcinoma, Carcinosarcoma with high grade serous or Grade 2/3 endometrioid components, or clear cell carcinoma (Pure or Mixed).
* Have measurable disease
* FRα-positive tumor expression as defined in the protocol
* Have at least one "target lesion" to be used to assess response as defined by RECIST v1.1
* Patients must have received prior treatment with ≤ 3 prior lines of therapy for recurrent disease; hormonal agents are not considered a line of therapy; prior treatment with folate receptor-targeting investigational agents is not allowed
* Have Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Time from prior therapy: Systemic anti-neoplastic therapy: five half-lives or four weeks, whichever is shorter; Radiotherapy: wide-field radiotherapy completed at least four weeks, or focal radiation completed at least two weeks, prior to starting study treatment
* Patients must have resolution of toxic effect(s) of the most recent prior chemotherapy
* Patients must have adequate hematologic, liver and kidney function as defined in the protocol
* Women of child bearing potential (WCBP), must agree to use effective contraceptive methods during study treatment and for at least twelve weeks after the last dose of IMGN853
* WCBP must have a negative pregnancy test within 4 days prior to the first dose of study treatment
* At time of initial surgery, patient may have either been optimally or suboptimally debulked
* Have signed the informed consent form, and willing to adhere to the study visit schedule and other protocol requirements
* ≥ 18 years of age

Exclusion Criteria:

* Active or chronic corneal disorder
* Serious concurrent illness or clinically-relevant active infection as defined in the protocol
* Clinically-significant cardiac disease such as recent myocardial infarction (≤ 6 months prior to day 1), unstable angina pectoris, uncontrolled congestive heart failure, uncontrolled hypertension, prior history of hypertensive crisis or hypertensive encephalopathy, uncontrolled cardiac arrhythmias, clinically-significant vascular disease, severe aortic stenosis, clinically significant peripheral vascular disease, or cardiac toxicity following prior chemotherapy
* History of neurological conditions
* History of hemorrhagic or ischemic stroke within the last 6 months
* History of cirrhotic liver disease
* Previous clinical diagnosis of non-infectious pneumonitis
* Prior hypersensitivity to monoclonal antibodies
* Women who are pregnant or breast feeding
* Carcinomatous meningitis, untreated central nervous system (CNS) disease or symptomatic CNS metastasis
* History or evidence of thrombotic or hemorrhagic disorders within 6 months before first study treatment
* Required used of folate-containing supplements (e.g. folate deficiency)
* Has a known additional malignancy that is progressing or required active treatment within 3 years of first dose of study treatment

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2020-07-15 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 5 Years
  Objective response rate (complete response and partial response rates) by RECIST 1.1 criteria of mirvetuximab soravtansine in patients with folate receptor α-positive persistent or recurrent endometrial cancer

SECONDARY OUTCOMES:
Duration of overall survival (OS) | 5 Years
  Overall survival is defined as the duration of time from study entry to time of death or the date of last contact.
Duration of progression free survival (PFS) | 5 Years
  Progression-free survival is defined as the duration of time from study entry to time of progression, death, or the date of last contact, whichever occurs first.
Durable disease control rate (DDCR) | 5 Years
  The percentage of patients who have achieved complete response, partial response, and stable disease.
Safety profile of mirvetuximab soravtansine (IMGN853) in endometrial cancer patients (adverse events as assessed by CTCAE v5.0) | 5 Years
  Incidence of treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro D. Santin, M.D., Principal Investigator — Yale University
Locations (1):
- Smilow Cancer Hospital at Yale New Haven, New Haven, Connecticut, United States